CLINICAL TRIAL: NCT03627468
Title: A Multicenter, Randomized, Open-label, Phase 3 Long-term Safety Study of Topically Applied Sofpironium Bromide (BBI-4000) Gel, 5% and 15% in Subjects With Axillary Hyperhidrosis
Brief Title: A Safety Study of BBI-4000 Gel in Patients With Axillary Hyperhidrosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Botanix Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BBI-4000-CL-303
Record Dates: First submitted 2018-08-02; First posted 2018-08-13 (Actual); Results first posted 2023-05-19 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-04

CONDITIONS: Primary Axillary Hyperhidrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Gel, 5% (Experimental): Sofpironium Bromide Gel, 5%, applied topically to each axilla once daily for 48 weeks
  Interventions: Drug: Sofpironium Bromide Gel, 5%
- Gel, 15% (Experimental): Sofpironium Bromide Gel, 15%, applied topically to each axilla once daily for 48 weeks
  Interventions: Drug: Sofpironium Bromide Gel, 15%

INTERVENTIONS:
Drug: Sofpironium Bromide Gel, 5% — Sofpironium Bromide Gel, 5%
  Other Names: BBI-4000
  Arms: Gel, 5%
Drug: Sofpironium Bromide Gel, 15% — Sofpironium Bromide Gel, 15%
  Other Names: BBI-4000
  Arms: Gel, 15%

SUMMARY:
Hyperhidrosis is a disorder of abnormal excessive sweating. Primary hyperhidrosis (armpits, hands, and feet) affects approximately 4.8% of the US population and is believed to be caused by an overactive cholinergic response of the sweat glands. Current therapies have limited effectiveness, significant side effects, and can be invasive and costly. Sofpironium bromide (BBI-4000) is a novel soft-drug in development for the topical treatment of hyperhidrosis. This Phase 3 study will assess the long-term safety, tolerability, and efficacy of sofpironium bromide gel applied topically to subjects with axillary hyperhidrosis.

DETAILED DESCRIPTION:
This is a randomized, open-label, phase 3 long-term study designed to evaluate the safety, local tolerability and efficacy of sofpironium bromide gel when applied topically to the axillae.

Subjects will apply the gel once daily at bedtime, to both axillae.

A maximum of 300 subjects, will be randomized to receive one of two sofpironium bromide gel concentrations.

Adverse events, vital signs, and local tolerability assessments will be collected at each visit. Urine pregnancy tests will be taken throughout the course of the study for women of child bearing potential. Blood and urine samples will be collected and analyzed for routine hematology, chemistry, and urinalysis parameters at specified visits. Patient-reported outcome assessments will be recorded during the study at predefined time points.

The study will be comprised of a total of 17 scheduled visits to take place over a 52 week period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject ≥9 years of age in good general health.
* Diagnosis of primary axillary hyperhidrosis that meets all the following criteria: (a) HDSM-Ax of 3 - 4 inclusive at both the Screening Visit (Visit 1) and Baseline Visit (Visit 2). (b) Symptoms of axillary hyperhidrosis for greater than or equal to 6 months' duration prior to Baseline Visit (Visit 2).

Exclusion Criteria:

* In the Investigator's opinion, any skin or subcutaneous tissue conditions of the axilla(e), (i.e., the axillary area should be deemed otherwise "normal", besides the hyperhidrosis diagnosis, and free of blisters, large boils or sinus tracts, significant scarring or open wounds).
* Prior use of any prohibited medication(s) or procedure(s) within the specified timeframe for the treatment of axillary hyperhidrosis: (a) Botulinum toxin to the axillary area within 6 months of the Baseline Visit (Visit 2). (b) Axillary thermolysis, sympathectomy or surgical procedures of the axillary area at any time in the past. (c) Serotonergic agonist (or drugs that increase serotonin activity including SSRIs), beta-blocker, alpha-adrenergic agonist (clonidine), dopamine partial agonist or tricyclic antidepressant treatment within 28 days of the Baseline Visit (Visit 2). However, if a subject has been on a stable dose (in the opinion of the PI) of any of these medications and has not had a recent change in hyperhidrosis frequency or severity for 3 months prior to the Baseline Visit; they may be included. Doses of these agents should not be altered during the course of the study. (d) Any topical treatment for hyperhidrosis, requiring a prescription, within 15 days of Baseline Visit (Visit 2).
* Anticholinergic agents used to treat conditions such as, but not limited to, hyperhidrosis, asthma, incontinence, gastrointestinal cramps, and muscular spasms by any route of administration (e.g., IV, oral, inhaled, topical) within 28 days of the Baseline Visit (Visit 2).
* Use of potent oral inhibitors of cytochrome P450 CYP3A & CYP2D6 and transporter inhibitors (OCT2/MATE1/MATE2) 14 days prior to the Baseline Visit (Visit 2). The use of topical antifungal medications is permitted if not applied in the treatment area.
* Any oral or topical homeopathic or herbal treatment (i.e., alternative therapies such as sage tablets, chamomile, valerian root and St. John's Wort) within 7 days of the Baseline Visit (Visit 2).
* Use of any cholinergic drug (e.g., bethanechol) within 15 days of the Baseline Visit (Visit 2).
* Use of any anti-anxiety and/or anti-depressant, amphetamine product or drugs with known anticholinergic side effects is prohibited with the following exceptions: (a) If a subject has been on a stable dose of an anti-anxiety and/or anti-depressant drug and has not had a recent change in hyperhidrosis frequency or severity for 3 months; they may be included. (b) An amphetamine product may be allowed if the dose has been stable for greater than or equal to 6 months without change in hyperhidrosis frequency or severity. (c) Drugs with known anticholinergic side effects (taken within the last 28 days), including dry mouth, blurred vision, may be allowed based on the Principal Investigator's assessment.

NOTE: If anticholinergic side effect(s) are experienced on these medications prior to starting study medication; document the side effect(s) and severities in the source document and the eCRF. The doses of these agents should not be altered during the course of the study.

* Known causes of hyperhidrosis or known history of a condition that may cause hyperhidrosis (i.e., hyperhidrosis secondary to any known cause such hyperthyroidism, diabetes mellitus, medications, etc.).
* Subjects with hyperhidrosis symptoms initiated or exacerbated with menopause.
* Subjects with unstable type 1 or type 2 diabetes mellitus or thyroid disease, history of renal impairment, hepatic impairment, malignancy, glaucoma, intestinal obstructive or motility disease, obstructive uropathy, myasthenia gravis, benign prostatic hyperplasia (BPH), neurological conditions, psychiatric conditions, Sjögren's syndrome, Sicca syndrome, or cardiac abnormalities that may alter normal sweat production or may be exacerbated by the use of anticholinergics in the Investigator's opinion.
* Known hypersensitivity to glycopyrrolate, anticholinergics, or any of the components of the topical formulation.
* Subject is pregnant, lactating or is planning to become pregnant during the study.
* Participating in a study of or used an investigational drug or device within 28 days prior to the Baseline Visit (Visit 2).
* Any major illness within 28 days before the screening examination.
* Any other condition, including psychiatric illness (depression and/or anxiety) that would interfere with study participation and/or evaluation of study endpoints or laboratory abnormality that, in the opinion of the Investigator, would put the subject at unacceptable risk for participation in the study or may interfere with the assessments included in the study.
* History or presence of supraventricular tachycardia, ventricular arrhythmias, atrial fibrillation or atrial flutter.

Ages: 9 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2020-01-27 (Actual); Study Completion 2020-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Walker, MD PhD, Study Director — Botanix Pharmaceuticals
Locations (12):
- United States (12):
  - Coastal Clinical Research, Inc., Mobile, Alabama
  - Northwest Arkansas Clinical Trials Center, Rogers, Arkansas
  - Center for Clinical and Cosmetic Research, Aventura, Florida
  - Skin Care Research, Inc., Boca Raton, Florida
  - Baumann Cosmetic & Research Institute, Miami, Florida
  - Tory Sullivan MD PA, North Miami Beach, Florida
  - Research Institute of the Southeast, LLC, West Palm Beach, Florida
  - Grekin Skin Institute, Warren, Michigan
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Tennessee Clinical Research Center, Nashville, Tennessee
  - J&S Studies, Inc., College Station, Texas
  - Austin Institute for Clinical Research, Pflugerville, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Gel, 5% | Gel, 15%
Started | 103 | 197
Completed | 72 | 118
Not Completed | 31 | 79
Not completed — Adverse Event | 5 | 33
Not completed — Withdrawal by Subject | 13 | 23
Not completed — Physician Decision | 1 | 0
Not completed — Protocol Violation | 0 | 2
Not completed — Lost to Follow-up | 10 | 16
Not completed — Death | 1 | 0
Not completed — Pregnancy | 1 | 1
Not completed — Lack of Efficacy | 0 | 2
Not completed — Poor Compliance or Noncompliance | 0 | 2

BASELINE CHARACTERISTICS:
Population: Population: Intent-to-Treat
Groups:
- Total: Total of all reporting groups
Arm/Group | Gel, 5% | Gel, 15% | Total
Number analyzed (Participants) | 103 | 197 | 300
Age, Customized [Count of Participants; unit: Participants]
  9-12 years | 1 | 0 | 1
  13-16 years | 3 | 14 | 17
  ≥17 years | 99 | 183 | 282
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 121 | 180
  Male | 44 | 76 | 120
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 39 | 65
  Not Hispanic or Latino | 76 | 157 | 233
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 4 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 28 | 47 | 75
  White | 74 | 143 | 217
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
HDSM-Ax-11 Scale Score Summary - Baseline Visit [Mean (Standard Deviation); unit: units on a scale] — HDSM-Ax-11:
  2/11 questions measure frequency underarm sweating. Responses: None of the time (0); A little of the time (1); Some of the time (2); Most of the time (3); All of the time (4) 7/11 questions measure severity underarm sweating. Responses: I did not experience this (0); Mild (1); Moderate (2); Severe (3); Very Severe (4).
  2/11 questions measure the need to change/clean from underarm sweating. Responses: Not at all (0); Slight (1); Moderate (2); Strong (3); Very Strong (4).
  Baseline individual mean scores calculated = the total numeric score / number of questions answered
  units on a scale | 3.57 (0.308) | 3.56 (0.316) | 3.565 (0.312)

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With Treatment Emergent Adverse Events Cumulative to Week 48 by Maximum Severity
Description: The number of participants with treatment emergent adverse events cumulative to week 48 by maximum severity based on a 3 point increasing severity scale of: mild, moderate and severe
Time Frame: All safety subjects, reaching week 48 or not
Population: Overall number of participants analyzed included the Safety Population. Subunits: Subjects reporting any TEAE made up the overall number of units analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Gel, 5% | Gel, 15%
Number analyzed (Participants) | 102 | 197
Participants
  Mild Severity | 27 | 55
  Moderate Severity | 29 | 58
  Severe Severity | 2 | 17
  Missing | 0 | 0
  No TEAE Reported | 44 | 67

2. Primary Outcome: Number of Participants With Post-baseline Local Tolerability Assessments Results by Treatment Group (Population: Safety)
Description: Number of participants reporting: local tolerability symptoms and severity (worst) symptom ratings; Incidence by subject report of any local symptom type (including Burning, Stinging, Itching, Scaling, Erythema) and local symptom worst severity rated either as Absent or Minimal, Mild, Moderate or Severe.
Time Frame: All Safety Subject, Baseline-Through study completion (48 weeks) or Not
Population: Safety population, units analyzed: subject incidence of report of any local symptom type (including Burning, Stinging, Itching, Scaling, Erythema) and local symptom worst severity rating either as Absent or Minimal, Mild, Moderate or Severe. Subjects where local tolerability assessment was not completed were also included.
Measure: Number; unit: participants
Arm/Group | Gel, 5% | Gel, 15%
Number analyzed (Participants) | 102 | 197
participants
  Absent | 31 | 59
  Minimal | 34 | 41
  Mild | 20 | 37
  Moderate | 12 | 38
  Severe | 4 | 19
  Subject Tolerability Assessment not Performed | 1 | 3

3. Secondary Outcome: The Number (%) of Subjects Achieving (-) ≥ 1point (Negative) Change (or Decrease) in the Hyperhidrosis Disease Severity Measure-Axillary 11-item (HDSM-Ax-11©) Score
Description: HDSM-Ax-11 is 11-question tool used to measure effect of BBI-4000 gel, 5% and 15 % on disease in subjects with axillary hyperhidrosis. Two questions measured frequency (since yesterday) of underarm sweating outcomes. The range of responses included increasing frequency scale: None of the time (0); A little of the time (1); Some of the time (2); Most of the time (3); All of the time (4). The next seven questions measured severity of underarm sweating outcomes. Range in increasing severity: I did not experience this (0); Mild (1); Moderate (2); Severe (3); Very Severe (4). The last two questions measured the need to change or clean from underarm sweating. Range in increasing degree of need: Not at all (0); Slight (1); Moderate (2); Strong (3); Very Strong (4).
  The individual mean was derived by taking the total score and dividing by the number of questions answered. A negative change (difference of mean HDSM-Ax-11total scores) reflected improvement in HDSM-Ax-11© score and condition.
Time Frame: From baseline to each visit through study completion (48 weeks)
Population: ITT population and subjects with Baseline-End of Treatment HDSM-Ax-11© scores
Measure: Count of Participants; unit: Participants
Arm/Group | Gel, 5% | Gel, 15%
Number analyzed (Participants) | 72 | 113
Participants
  Observed ≥1- point HDSM-AX-11 decrease: YES | 61 | 95
  Observed ≥1- point HDSM-AX-11 decrease: NO | 11 | 18

4. Secondary Outcome: The Number (%) of Subjects Achieving (-) ≥ 1.5 Point (Negative) Change (or Decrease) in the Hyperhidrosis Disease Severity Measure-Axillary 11-item (HDSM-Ax-11©) Score
Description: HDSM-Ax-11 is 11-question tool used to measure effect of BBI-4000 gel, 5% and 15 % on disease in subjects with axillary hyperhidrosis. Two questions measured the frequency (since yesterday) of underarm sweating outcomes. The range of responses included increasing frequency scale: None of the time (0); A little of the time (1); Some of the time (2); Most of the time (3); All of the time (4). The next seven questions measured the severity of underarm sweating outcomes. Range in increasing severity: I did not experience this (0); Mild (1); Moderate (2); Severe (3); Very Severe (4). The last two questions measured the need to change or clean from underarm sweating. Range in increasing degree of need: Not at all (0); Slight (1); Moderate (2); Strong (3); Very Strong (4).
  The individual mean was derived by taking the total score and dividing by the number of questions answered. A negative change (difference of mean HDSM-Ax-11scores) reflected improvement in HDSM-Ax-11© score and condition.
Time Frame: From baseline to each visit through study completion (48 weeks)
Population: ITT population and subjects with Baseline-End of Treatment HDSM-Ax-11© scores
Measure: Count of Participants; unit: Participants
Arm/Group | Gel, 5% | Gel, 15%
Number analyzed (Participants) | 72 | 113
Participants
  Observed ≥1.5 - point HDSM-AX-11 decrease: YES | 55 | 80
  Observed ≥1.5 - point HDSM-AX-11 decrease: NO | 17 | 33

5. Secondary Outcome: The Number (%) of Subjects Achieving (-) ≥ 2 Point (Negative) Change (or Decrease) in the Hyperhidrosis Disease Severity Measure-Axillary 11-item (HDSM-Ax-11©) Score
Description: as for outcome 4
Time Frame: From baseline to each visit through study completion (48 weeks)
Population: ITT population and subjects with Baseline-End of Treatment HDSM-Ax-11© scores
Measure: Count of Participants; unit: Participants
Arm/Group | Gel, 5% | Gel, 15%
Number analyzed (Participants) | 72 | 113
Participants
  Observed ≥2- point HDSM-AX-11 decrease: YES | 51 | 70
  Observed ≥2- point HDSM-AX-11 decrease: NO | 21 | 43

ADVERSE EVENTS:
Time Frame: Each Subject's AE data was collected over approximately 52 weeks of participation, including 48 weeks of investigational treatment.
Arm/Group | Gel, 5% | Gel, 15%
All-Cause Mortality (participants affected / at risk) | 1/102 | 0/197
Serious Adverse Events (participants affected / at risk) | 1/102 | 4/197
Other Adverse Events (participants affected / at risk) | 58/102 | 131/197
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gel, 5% (N=102) | Gel, 15% (N=197)
Depression (Psychiatric disorders) | 0 | 1
Suicide Attempt (Psychiatric disorders) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Septic Shock (Infections and infestations) | 1 | 0
Cardiac Myxoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Gel, 5% (N=102) | Gel, 15% (N=197)
Application site pruritus (General disorders) | 6 | 29
Application site pain (General disorders) | 4 | 29
Application site dermatitis (General disorders) | 6 | 21
Application site erythema (General disorders) | 6 | 15
Application site irritation (General disorders) | 5 | 11
Application site rash (General disorders) | 1 | 8
Application site exfoliation (General disorders) | 2 | 6
Application site dryness (General disorders) | 0 | 4
Upper respiratory tract infection (Infections and infestations) | 9 | 8
Nasopharyngitis (Infections and infestations) | 5 | 3
Viral upper respiratory tract infection (Infections and infestations) | 4 | 4
Influenza (Infections and infestations) | 2 | 4
Application site folliculitis (Infections and infestations) | 0 | 5
Pneumonia (Infections and infestations) | 3 | 0
Dry Mouth (Gastrointestinal disorders) | 9 | 33
Vision Blurred (Eye disorders) | 5 | 37
Mydriasis (Eye disorders) | 1 | 10
Dry eye (Eye disorders) | 1 | 7
Urinary retention (Renal and urinary disorders) | 3 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 0
Headache (Nervous system disorders) | 1 | 4
Hypertension (Vascular disorders) | 1 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Agreement terms prioritized a multi-center publication at the study end. Should such a publication not be completed, an investigator right to individually publish results of his/her study (limited to his/her site data) was included, if for purely scientific or educational purposes; not for any commercial purposes. PI(s) were to submit draft materials to the Sponsor 60 days prior to Investigator release of individual abstract or manuscript. Additional disclosure restrictions and terms applied .

DOCUMENTS (2):
  • Study Protocol (2018-05-15): https://cdn.clinicaltrials.gov/large-docs/68/NCT03627468/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-24): https://cdn.clinicaltrials.gov/large-docs/68/NCT03627468/SAP_001.pdf